CLINICAL TRIAL: NCT02435186
Title: Recombinant Adenoviral p53 Human Gene Combined With Chemotherapy in Treatment of Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, and Primary Peritoneal Cancer
Brief Title: p53 Gene in Treatment of Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, and Primary Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rAd-p53-H20150111
Record Dates: First submitted 2015-04-28; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Ovarian Epithelial Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: p53 gene; chemotherapy; recurrent; epithelial; ovarian cancer; fallopian tube cancer; primary peritoneal cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Recurrence; Ovarian Neoplasms | interventions — Genes, p53; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- p53 gene plus chemotherapy (Experimental): Intraperitoneal p53 gene plus cisplatin, and paclitaxel iv
  Interventions: Drug: p53 gene; Drug: Cisplatin; Drug: Paclitaxel
- chemotherapy (Active Comparator): Intraperitoneal cisplatin, and paclitaxel iv
  Interventions: Drug: Cisplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: p53 gene — p53 gene will be given intraperitoneally.
  Other Names: recombinant adenoviral human p53 gene
  Arms: p53 gene plus chemotherapy
Drug: Cisplatin — 150 mg/m^2 cisplatin will be given intraperitoneally.
Drug: Paclitaxel — Paclitaxel (175 mg/m2, 3 h) will be given by iv

SUMMARY:
The study objective is to investigate the efficacy and safety of p53 combined with chemotherapy (cisplatin and paclitaxel) in treatment of recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, and Primary Peritoneal Cancer.

DETAILED DESCRIPTION:
The study objective is to investigate the efficacy and safety of p53 combined with chemotherapy (cisplatin and paclitaxel) in treatment of recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, and Primary Peritoneal Cancer.

study design: open-labeled, active controlled, randomized, phase 2 treatments: experiment group will consist of intraperitoneal p53 (2 x 10^12 viral particles) plus cisplatin 150 mg/m^2, and Paclitaxel 175 mg/m^2 IV over 3 h on day 1; every 21 d for 6 cycles.

study end points: response rate, progression-free survival, overall survival and Karnofsky score（KPS).

ELIGIBILITY:
Inclusion Criteria:

1. histopathologically diagnosed ovarian epithelial cancer, fallopian tube cancer, and primary peritoneal cancer
2. recurrent
3. 18 years or older
4. with normal tests of hemogram, blood coagulation, liver and kidney function
5. signed the informed consent form.

Exclusion Criteria:

1. Serious blood coagulation disorder, bleeding tendency, platelet < 6 * 1000000000/L;
2. have serious heart, lung function abnormalities or severe diabetes patients;
3. active infection;
4. severe atherosclerosis;
5. AIDS patients;
6. serious thrombotic or embolic events within 6 months;
7. renal insufficiency requiring hemodialysis or peritoneal dialysis;
8. pregnant or lactating women;
9. mental disorder or disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
response rate | from starting study treatment to 6 months
  Objective response rate using RECIST version 1.1 guidance
progress-free survival | from starting treatment to 2 years after
  measure the time to progression/death, or to the last tumor assessment

SECONDARY OUTCOMES:
overall survival | from starting study treatment to 2 years after
  measure the time to death, or time last known alive
Karnofsky Performance Status score（KPS） | from starting study treatment to 2 years after
safety as measured by adverse events, vital signs, clinical lab tests, ECG and physical examination | from starting study treatment to 30 days after the last study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- xijing hospital in China Medical University, Shenyang, Liaoning, China